CLINICAL TRIAL: NCT03404440
Title: Eradication of Helicobacter Pylori With a Lactobacillus Reuteri Strain Combination (Strains DSM 17938 and ATCC PTA 6475) and a Proton Pump Inhibitor
Brief Title: Eradication of Helicobacter Pylori With a Lactobacillus Reuteri Strain Plus Proton Pump Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LRHPPPI
Record Dates: First submitted 2017-12-30; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori; L. Reuteri; Proton Pump Inhibitor

STUDY DESIGN:
Intervention Model Description: double-blind randomized, parallel-group, placebo-controlled study.
Who Masked: Participant, Investigator
Masking Description: Placebo capsules were identical in shape, colour and taste to Gastrus capsules but without L. reuteri
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L.Reuteri (Active Comparator): Lactobacillus reuteri DSM 17938 + Lactobacillus reuteri ATCC PTA 6475 one tablet by mouth 7 times per day + Pantoprazole 20 mg twice a day for 28 days
  Interventions: Other: L.Reuteri
- Placebo (Placebo Comparator): Placebo one tablet by mouth 7 times per day + Pantoprazole 20 mg twice a day for 28 days
  Interventions: Other: L.Reuteri

INTERVENTIONS:
Other: L.Reuteri
  Other Names: Gastrus

SUMMARY:
Meta-analyses involving >4000 subjects with probiotics added to antimicrobial Helicobacter pylori eradication therapy in populations with antibiotic resistance have reported a mean increase in eradication rate of 12.2%. It is unclear how to translate that result into clinical practice.

To evaluate whether administration of Lactobacillus reuteri plus a PPI without antibiotics would eradicate H. pylori infections.

This was a double-blind placebo-controlled randomized 2 site study of L. reuteri (2 x 108 CFU L. reuteri DSM 17938 plus 2 x 108 CFU L. reuteri ATCC PTA 6475) 7 times per day or matching placebo plus 20 mg pantoprazole b.i.d. for 4 weeks. Cure was defined by negative 13C-UBT, 4 weeks after therapy. Sample size was based on obtaining >50% cures to be clinically useful as monotherapy.

DETAILED DESCRIPTION:
Aim of study This double-blind study will assess if the combination of PPI and a strain combination (Gastrus) of L.reuteri can yield higher eradication rates if doses are increased and dose interval shortened. The aim is to achieve at least 50% eradication as assessed by UBT.

Study Product

Gastrus capsules:

2x108 CFU Lactobacillus reuteri DSM 17938 + 2x108 CFU Lactobacillus reuteri ATCC PTA 6475.

Placebo capsules:

Identical in shape, colour and taste to Gastrus capsules but without the Lactobacillus reuteri components.

Both study products are delivered in identical containers containing 30 capsules.

Dosing Group 1: 1 Gastrus capsule 7 times per day + Pantoprazole 20 mg b.i.d. Group 2: 1 placebo capsule 7 times per day + Pantoprazole 20 mg b.i.d. One capsule of the Study Product are to be taken every 2-3 hours 7 times per day.

The Study Product containers will be collected at the day 28 visit and remaining tablets are counted and compliance checked.

40 mg Pantoprazole is to be taken just before breakfast and dinner (i.e. daily dose 80 mg).

Length of treatment The optimal length of dosing needed is unknown. Saggioro and Francavilla used 30 and 28 days respectively and Dore et al had a 60-day regimen. From a practical/economical/tolerability point of view, a 28-day regimen is suggested in order to shorten the time to triple-therapy for those non-eradicated. Those patients with H. pylori at the second UBT/Endoscopy (i.e. treatment failures) will be offered standard eradication therapy.

Compliance, PP and ITT In order to be assessed as "compliant" the participant should have consumed at least 75% (or other?) of the allotted doses. In order to improve compliance, the participants will be equipped with alarm-devices. Compliant patients will be assessed as Per-Protocol (PP). Patients that are non-compliant but have consumed at least one full day of doses (i.e. 14 tablets) will be included in the Intention-To-Treat analysis.

Outcomes Primary efficacy parameter Number of H. pylori-eradicated at 9 weeks as evidenced by Δ-13C-UBT < 5 ppm. The difference between active and placebo treatment will be compared.

Exploratory parameters Changes in GSRS at 4 and 9 weeks as compared to baseline and between groups. Changes of the gastric microbiota in the presence of PPI with or without Gastrus.

Sample size calculation Assuming that the spontaneous eradication is 5% or less, and that the desired eradication rate on active treatment is >50%, 23 subjects are needed in each group with a power of 90% and a confidence level of 95%. To correct for potential drop-outs, 25 subjects will be recruited to each group.

Ethical committee The study protocol will have to be approved by the local ethical committee before study start. Once approved, a protocol summary will be posted on clinicaltrials.gov.

Study flow and procedures Randomisation & labelling Randomisation will be computerised using the tool provided by randomizer.org. A third party not otherwise involved in the study will label active and placebo Study Product. Randomisation lists will be kept in sealed envelopes at the study sites and a sealed copy will also be kept at BioGaia. The envelopes may not be open until all study data have been entered into the database and until the database has been locked. However, see "Serious Adverse Event" below.

Patients will be entered into the study sequentially by allocating the lowest available remaining randomisation number to the patient.

Procedures Histology During endoscopy two biopsy specimens are taken from the antrum, one from the angulus and two from the corpus. Hp-infection is defined as the presence of typical histology and bacteria on histological examination of biopsies stained by H&E and GIEMSA. One additional biopsy from the corpus area is placed in PBS with 5% glycerol and stored at - 70 oC until further processing for microbiota analyses (see below.

Gastric microbiota analysis Bacterial DNA extraction and sequencing for microbiota analyses is performed according to a standardised protocol (Willing BP et. al 2010). Analysis of community structure focuses on sequencing of targeted regions e.g. the 16S rRNA gene using the Illumina Miseq high-throughput sequencing platform. Sequences are finally processed with the QIIME 1.8.0 pipeline (Caporaso JG et. al 2010).

13C-UBT According to standard protocol (Gatta L., et al. 2006). After the first UBT needed for inclusion, a second UBT will be performed at 8-9 weeks (4-5 weeks after end of study treatment) to assess Hp status.

Gastrointestinal Symptom Rating Scale (GSRS). Participants will be asked to fill out the GSRS questionnaire after inclusion but before taking the first dose of study product, at 4 weeks (end of treatment) and at 8-9 weeks (at follow-up UBT) (Svedlund J. et al. 1988) Data collection The Principal Investigator will prepare one set of Case Record Forms (CRF) for each patient in which all data pertinent to the study will be entered.

Statistical methods All efficacy parameters will be analysed according to both ITT and PP. Safety considerations The investigator is responsible for monitoring the safety of subjects who have entered the study. All adverse events (AE) occurring after any administration of the study product will be followed to the end of the study or until resolution. AE will be evaluated by the Investigator and reported in the CRF.

Serious adverse events, as defined below, must be reported to the sponsor within 24 hours of when the investigator became aware of the SAE. It is also important to report all adverse events that result in permanent discontinuation of the study product, whether serious or non-serious.

Adverse Events An adverse event (AE) is any undesirable medical occurrence in a subject administered a study product, regardless of causality assessment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study product, whether or not considered related to the study product. All adverse events, including observed or volunteered problems, complaints, or symptoms are to be recorded on the case report form (CRF). Each adverse event is to be evaluated for duration, intensity, and causal relationship with the study product or other factors.

Subjects should be instructed to report any AE that they experience to the Investigator. Investigators should assess for AE at each visit. AE occurring during the clinical trial, including the follow-up period should be recorded on the appropriate AE CRF. To capture the most potentially relevant safety information during a clinical trial, it is important that investigators record accurate AE terms on CRF.

If discernible at the time of completing an AE in CRF, a specific disease or syndrome rather than individual associated signs and symptoms should be identified by the investigator and recorded on the CRF. However, if an observed or reported sign or symptom is not considered a component of a specific disease or syndrome by the investigator, it should be recorded as a separate AE on the CRF. Laboratory values will be collected on the laboratory CRF. Do not enter changes from baseline in laboratory values on the AE CRF.

Serious Adverse Events A serious adverse event (SAE) is any AE that results in death is immediately life threatening requires or prolongs hospitalisation results in persistent or significant disability/incapacity is a medically significant event for any reason. Breaking the randomisation code In case that the responsible investigator decides that the randomisation code has to be revealed because that the AE may have been caused by the Study Product and that un-blinding is of essence for the further treatment of the patient, the following procedure will be followed: The responsible investigator will assign a professional otherwise not involved in the study to un-blind the Study Product for the specific patient. He/she will open the sealed envelope, find the relevant randomisation number and inform the responsible investigator without revealing any other randomisation numbers. He/she will then re-seal the envelope with transparent tape, date and sign on the tape.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for upper endoscopy for any reason
* Biopsy specimens indicative of Hp infection
* 13C-UBT indicative of Hp infection
* > 18 years of age
* Informed consent obtained

Exclusion Criteria:

* Severe gastritis
* Peptic ulcer
* Pregnancy or lactation
* Malignancy
* Other clinically significant condition
* Alcohol abuse
* Drug abuse
* Patients taking bismuth compounds, anti-secretory drugs, antibiotics or probiotics during 4 weeks preceding endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Eradication | Four weeks after post treatmetn assessed by Δ-13C-UBT
  number of patients with H. pylori infection eradicated at 9 weeks assessed by Δ-13C-UBT <5‰

CONTACTS AND LOCATIONS:
Overall Officials: ruggiero francavilla, Md PhD, Principal Investigator — University of Bari
Locations (1):
- Clinica Pediatrica, Bari, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bibbo S, Ahlstrom G, Pes GM, Graham DY, Engstrand L, Merola E, Dore MP. Resilience of the Gut Microbiome to Short Proton Pump Inhibitor Therapy With or Without High-Dosage L. reuteri in H. pylori-Infected Adults. Helicobacter. 2025 Sep-Oct;30(5):e70064. doi: 10.1111/hel.70064. PMID 40993967
- [Derived] Dore MP, Bibbo S, Pes GM, Francavilla R, Graham DY. Role of Probiotics in Helicobacter pylori Eradication: Lessons from a Study of Lactobacillus reuteri Strains DSM 17938 and ATCC PTA 6475 (Gastrus(R)) and a Proton-Pump Inhibitor. Can J Infect Dis Med Microbiol. 2019 Apr 1;2019:3409820. doi: 10.1155/2019/3409820. eCollection 2019. PMID 31065301